CLINICAL TRIAL: NCT01481207
Title: Magnetic Resonance Imaging (MRI) and Spectroscopy (MRS) Biomarkers of Neonatal Hypoxic Ischemic Encephalopathy
Brief Title: Magnetic Resonance Imaging and Spectroscopy Biomarkers of Neonatal Hypoxic Ischemic Encephalopathy
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: CIV-11-11-002981
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: magnetic resonance spectroscopy; magnetic resonance imaging
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- neonates with perinatal asphyxia: neonates with suspected perinatal asphyxia (HIE)

SUMMARY:
Neonatal hypoxic ischemic encephalopathy (HIE) is a serious neurological condition characterised by acute or subacute brain injury arising from perinatal hypoxia. HIE is thought to affect approximately 0.2% of live births, and is associated with a high risk of mortality or long-term neurological disability.

Accurate biomarkers for long-term neuro-developmental outcome following HIE are extremely important both for clinical management and the evaluation of therapeutic approaches. According to a recent meta-analysis, the ratio of the cerebral concentrations of lactate and N-acetyl aspartate (NAA), two neuro-metabolites detectable with magnetic resonance spectroscopy (MRS), currently represents the most accurate prognostic indicator of outcome following HIE. However, for various technical reasons standard MRS methods do not offer optimal sensitivity for detecting lactate, which may potentially be improved with a custom lactate editing MRS sequence. In addition, while perfusion has also been suggested as a potential biomarker for neuro-developmental outcome following HIE, due to a paucity of MR perfusion imaging studies in neonates, the prognostic accuracy of perfusion MR measures has not been evaluated in comparison with more established MR biomarkers. The aims of this study are:

1. to evaluate the relative sensitivity of a custom lactate editing MRS pulse sequence (specialist software) relative to the standard point resolved (PRESS) MRS sequence for detecting lactate in neonates with suspected HIE.
2. to evaluate the sensitivity and specificity of MR perfusion measures in comparison to MRS measures as predictors of neuro-developmental outcome at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants (born at >36 weeks) with suspected perinatal asphyxia. Written informed consent from both parents.

Exclusion Criteria:

* Prematurity (born at < 36 weeks). Lack of written informed consent from both parents.

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates with suspected hypoxic ischemic encephalopathy
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-09; Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
sensitivity of lactate editing MR spectroscopy sequence (software) relative to that of the standard MR spectroscopy sequence. | 12 months
  The primary end-point will be reached when lactate and perfusion data have been collected from 30 neonates. The efficacy of the custom-MRS lactate editing sequence will be assessed relative to that of the standard MRS sequence for the detection of lactate (by comparing the lactate concentration (in mM) measured from the lactate edited MR spectra to that measured from the standard MR spectra).

SECONDARY OUTCOMES:
prognostic accuracy (sensitivity and specificity) of MRI and MRS for predicting motor outcome at age 2 | 3 years
  The secondary end-point will be reached upon completion of a neurological development assessment at the age of 2 years. Patients will be classified as having a good or poor outcome based on their motor skills at age 2, and the prognostic accuracy (eg sensitivity and specificity for predicting neuromotor outcome) of the standard and new MRI and MRS sequences will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth L O'Gorman, phD, Principal Investigator — University Children's Hospital Zurich, MRI Center
Locations (1):
- University Children's Hospital Zurich, MRI Center, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No